CLINICAL TRIAL: NCT01943149
Title: E-MAX 2nd Generation Vitamin E Polyethylene On BIOLOX Delta Ceramic Heads
Brief Title: E-MAX 2nd Gen Vit E Poly On BIOLOX Delta Ceramic Heads
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Renovis Surgical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HIP-001
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: In Need of a Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to monitor outcomes of total hip arthroplasties performed with E-MAX polyethylene and BIOLOX Delta Ceramic head. Polyethylene has been used as a bearing surface in total joint replacements for half of a century. Radiation, the most common form of sterilization, unfortunately it results in the creation of free radicals (atoms or molecules that cause chemical reactions with other substances) within the materials which cause the breakdown of the polyethylene. Second generation antioxidant polyethylene, Renovis E-MAX, mechanically blends in Vitamin E as an antioxidant. This helps eliminate free radicals while maintaining mechanical strength. The theory is that E-MAX will be a safe and long lasting bearing surface in total hip arthroplasty that meets or exceeds current wear rates after being placed in a patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient is under 65 years of age
* Patient's health status qualifies as ASA 1 or ASA 2
* Patient is willing to commit to long term follow (study duration is 10 yrs)

Exclusion Criteria:

* Allergy to any materials used in hip implant
* Unwillingness to participate in long term follow-up
* Diagnosis of inflammatory arthritis
* Simultaneous bilateral total hip arthroplasty is recommended.
* Patient's health status qualifies as ASA 3 or greater.
* Patient is over the age of 65 of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be patients of specified doctors specialized in orthopedic medicine with a specialty in joint replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
E-Max liner wear rate | Change from baseline to 10 years post-operative
  This measure's purpose it to look at the longevity of our product. Radiographs will be taken at standard checkpoints over the course of 10 years. Radiographic analysis will be done to assess wear rates of the E-Max liner over the course of the 10 year study. Wear rates will then be compared to other products that have already been studied and published in hopes of finding that E-Max's wear rates are at least as good if not better than comparative products on the market.

SECONDARY OUTCOMES:
Patient Function and Mobility | Change from Pre-operative to 10 years post-operative
  This measure will assess patient function and mobility preoperatively and compare this at standard checkpoints over 10 years post-operatively. This will be done through use of the Harris Hip Score and UCLA Functional Assessment with the hope of seeing improvement in both over the course of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornerstone Orthopedics, Louisville, Colorado, United States